CLINICAL TRIAL: NCT02553954
Title: Molecular Mechanisms of Senescence Predisposing to Cancer : Exploratory Analysis on Healthy Tissues Collected for Two Age Groups.
Brief Title: Molecular Mechanisms of Senescence Predisposing to Cancer : Exploratory Analysis on Healthy Tissues (SkinAge).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Oscar Lambret (Other)
Collaborators: Institut de Biologie de Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SkinAge-1306; 2013-A01793-42 (Other: ANSM)
Record Dates: First submitted 2015-09-17; First posted 2015-09-18 (Estimated); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Sarcoma
Keywords: Mechanisms of Senescence; Senescence markers
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Collection of healthy skin tissue (Experimental): Collection of healthy skin tissue
  Interventions: Procedure: Collection of healthy skin tissue

INTERVENTIONS:
Procedure: Collection of healthy skin tissue — Collection of two samples of healthy skin tissue, without disfigurement, during an intervention under general anesthesia for the treatment of a benign or malignant tumor.

SUMMARY:
Epidemiological data show that the incidence of carcinoma, the most common cancer, is strongly linked to the age. Non Melanoma Skin Carcinomas (NMSCs) (the most frequent cancers in the elderly population) derive from keratinocytes of the basal layer of the epidermis, from differentiated keratinocytes of the more superficial layers or from stem cells of hair follicles. Unlike NMSCs, soft-tissue sarcomas, including those deriving from dermal fibroblasts, are very rare (less than 1% of all cancers). Our overall purpose is to decipher the molecular pathways activated during the aging of these tissues that may explain why they have a so different propensity to undergo a malignant transformation. Given that senescent cells accumulate in the dermis and epidermis with age, we will constitute two groups : "young skin" that we arbitrarily limit to the range ≥ 18 and ≤ 40 and "aged skin" ≥ 55.

Thus the main objective of our study is to search within 2 age groups (≥ 18 and ≤ 40 years and ≥ 55 years) the expression of senescence markers on healthy skin tissue.

DETAILED DESCRIPTION:
* Information and obtaining informed consent.
* Collection of clinical data.
* Collection of two samples of healthy skin tissue, without disfigurement, during an intervention under general anesthesia for the treatment of a sarcoma.
* Freezing samples of healthy skin tissue in liquid nitrogen within 10 minutes after collection.
* Transfer of the samples to the laboratory of anatomopathology.
* Preparation of the healthy skin samples by the laboratory of anatomopathology.
* Transfer of the conditioned samples to the Institut de Biologie de Lille for analysis.
* Control of the aesthetic appearance during the postoperative consultation.
* Destruction of the samples at the end of analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an operable sarcoma
* Requiring a surgical operation under general anesthesia at the Oscar Lambret Centre
* Age ≥ 18 ans, belonging to one of the two following age groups : [ ≥ 18 and ≤ 40 years] and [ ≥ 55 years]
* Patient having a social security scheme
* Patient having signed an informed consent form for the study

Exclusion Criteria:

* Patient aged under 18 or between 41 and 54
* Location of the tumor on the face, neck or neckline
* Patient with a skin tumor
* Tumor-induced cutaneous fistula making suspect a tumor invasion of the skin
* Patient with a chronic skin disease
* Collection in an area already treated by surgery, radiotherapy or brachytherapy
* Pregnant or breastfeeding women
* Patient under guardianship or tutorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-10-07 (Actual); Primary Completion 2019-04-16 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Expression of senescence markers in healthy skin tissues collected for the two age groups. | Baseline

SECONDARY OUTCOMES:
Research of emerging cells in the skin tissue of the subjects of the two age groups via the expression of the Protease-Activated Receptor-1 (PAR-1). | Baseline
Presence of different types of DNA damage (single and double strand breaks) in the keratinocytes and fibroblasts of the skin tissues of the two age groups. | Baseline
Morbidity | Baseline
  Postoperative complications up to 30 days after surgery according to the Clavien-Dindo classification (2009), according to the NCI-CTCAE v4.0 beyond this deadline.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas PENEL, MD, Study Chair — Centre Oscar Lambret; Olivier PLUQUET, Study Director — Institut de Biologie de Lille
Locations (1):
- Centre Oscar Lambret, Lille, France

IPD SHARING:
Plan to Share IPD: No